CLINICAL TRIAL: NCT00817310
Title: Influence of Altered Cerebral Spinal Fluid and Arterial Flows on Cerebral Processing Functions in Premature Infants With Severe Intraventricular Hemorrhage
Brief Title: Neurophysiology and Anatomy of Severe Intraventricular Hemorrhage (IVH)
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nathalie Maitre, Assistant Professor, Vanderbilt University
Other Study IDs: PEDNE4 ML9999 18185 04550
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Intracranial Hemorrhages; Prematurity
MeSH Terms: conditions — Intracranial Hemorrhages; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Severe IVH: Infants born at less than 1500g with diagnosis of Grade II or IV IVH
- control: infants born at less than 1500g without IVH on HUS

SUMMARY:
Currently, when premature infants develop severe intraventricular hemorrhage (IVH), a type of intracerebral bleed, there are no proven therapeutic interventions to prevent the devastating consequences of this event. These children will be likely to develop cerebral palsy or severe cognitive delays.

The purpose of our study is to characterize differences in brain physiology, imaging, and function between premature infants with severe IVH and controls. The goals for gathering this information are to generate baseline data, which could facilitate early screening for complications of IVH in premature infants. These baseline data would also allow the design and implementation of early therapeutic interventions to help rehabilitate premature infants with severe IVH.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1500 grams for all inborn infants and age less than 14 post-natal days
* Birth weight < 1500 grams for all outborn infants transferred to the VCH NICU within the first 72 hours after birth and age less than 14 post-natal days
* Parents agree to their infant's participation and give informed written consent.

Exclusion Criteria:

* Unable to obtain informed consent.
* Congenital brain malformations leading to hydrocephalus
* Genetic and metabolic disorders leading to cerebral pathology

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with birthweights below 1500g that are between 1 and 14 days of age
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
neurodevelopmental outcome | 3 years
  BSID III scores

CONTACTS AND LOCATIONS:
Locations (1):
- Monroe Carell Children's Hospital at Vanderbilt, NICU, Nashville, Tennessee, United States